CLINICAL TRIAL: NCT07343518
Title: Effects of Sulforaphane Supplementation on Athletic Performance: a Double-blinded Randomized Crossover Study
Brief Title: Effects of Sulforaphane Supplementation on Athletic Performance
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maia (Other)
Responsible Party: Principal Investigator, Filipe Silvano Pinto Maia, Principal Investigator, University of Maia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: SFN_001
Record Dates: First submitted 2025-12-20; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Nutrition; Sports
Keywords: sulforaphane; fatigue; athletic performance
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Both participants and investigator will be blinded to the experimental conditions. Both placebo and supplementation will have the same appearence. Only the outcome assessor will know the assigned sequence to each participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sulforaphane (Experimental): Sulforaphane supplementation (Nomio)
  Interventions: Other: Fatigue protocol
- Placebo (Placebo Comparator): Placebo intervention
  Interventions: Other: Fatigue protocol

INTERVENTIONS:
Other: Fatigue protocol — Fatigue protocol comprising 6 sets of 30 seconds at 120% of velocity of maximal oxygen consumption

SUMMARY:
Considering the promising effects observed and the scarce and incipient scientific background of SFN in sports, the present study aims to evaluate the effects of SFN supplementation on fatigue, EIMD and recovery in trained individuals. In particular, outcomes such as time to exhaustion (TTE), and perceptual questionnaires of muscle soreness, recovery, and fatigue will be assessed, aiming to explore the effectiveness of SFN.

ELIGIBILITY:
Inclusion Criteria:

* Physically active individuals (engaging in exercise 3 or more times per week)

Exclusion Criteria:

* Individuals that experience musculoskeletal injuries or have experienced in the past 3 months

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
time to exhaustion | 24 hours

SECONDARY OUTCOMES:
Rating of Fatigue Scale | Baseline, 30 minutes, 24 hours
Total Quality Recovery Scale | Baseline, 30 minutes, 24 hours
Muscle soreness (Visual analogue scale) | Baseline, 30 minutes, 24 hours
Rating of perceived exertion scale | 30 minutes

IPD SHARING:
Plan to Share IPD: Undecided